CLINICAL TRIAL: NCT04435873
Title: Assessing Patient-Reported Experience of Care for Home Dialysis (ASPIRED)
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: SP124 Home Experience
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-05

CONDITIONS: Home Dialysis; End Stage Renal Disease
Keywords: ESRD; Dialysis; Patient Experience; Home Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mail Survey Participants: Approximately 1200 home patients will receive mail surveys. Of these, one thousand and twenty (1,020) patients will be asked to complete the survey once. One hundred and eighty (180) patients will be asked to complete the survey twice.
  Interventions: Other: Survey using "Your Home Dialysis Care Experience" tool.
- Telephone Survey Participants: Three hundred (300) home patients will be surveyed by phone. Of those, one hundred and twenty will be asked to complete the survey once. One hundred and eighty patients will be asked to complete the phone surveys on two separate occasions.
  Interventions: Other: Survey using "Your Home Dialysis Care Experience" tool.

INTERVENTIONS:
Other: Survey using "Your Home Dialysis Care Experience" tool. — Validation of a new survey instrument to capture the experience of care by home dialysis patients.

SUMMARY:
Home dialysis modalities, including peritoneal dialysis (PD) and home hemodialysis (HHD), represent alternatives to conventional in-center hemodialysis (HD) that for some patients may be better aligned with preferences regarding the integration of dialysis treatments into their lives. Assessment of patient experience and satisfaction with care among individuals undergoing maintenance dialysis in the United States is a national health care priority and mandated by Congress. While validated instruments (ICH CAHPS) are in use to assess patient experience with in-center HD, currently no validated instruments are available to measure patient-reported experience in home dialysis.

This Home Patient Experience Survey Validation Study is an in-house research study conducted in partnership with the University of Washington.

DETAILED DESCRIPTION:
Assessment of patient experience and satisfaction with care among individuals undergoing maintenance dialysis in the United States is a national health care priority and mandated by Congress. No validated instruments are available to measure the patient-reported experience of care in-home dialysis patients. Such tools are needed as more patients are expected to choose home dialysis therapies in the future. This study aims to validate a home patient experience survey instrument.

This is a cross-sectional validation to determine the measurement properties of a new home dialysis patient experience survey instrument. Satellite Healthcare home dialysis patients will be approached by mail or by phone to complete the survey.

The aim of this study is to perform field testing for this newly developed instrument for the purposes of instrument validation and to determine survey instrument measurement properties. This will include the evaluation of any multi-item scales as well as an overall score.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving care for home dialysis at a facility that provides care for >= 3 patients at the time of cohort identification.

Exclusion Criteria:

* Age < 18 years
* Patients receiving care for home dialysis at the facility for less than 3 months
* Institutionalized (senior nursing facility/multi-resident facility) or Hospice care patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population is composed of those individuals receiving Home Dialysis care at Satellite Healthcare facilities,
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the measurement model | through survey completion, an average of 6 months
  The evaluation will encompass the survey burden, presence of a floor or ceiling effect for any item, test-retest reliability, development of multi-item subscales, internal consistency and reliability, center level reliability of the items and composites, and construct validity.

SECONDARY OUTCOMES:
Survey response rate | through survey completion, an average of 6 months
  Percent (%) of participants contacted who complete survey instrument

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Satellite WellBound of Daly City, Daly City, California
  - Satellite Wellbound of Emeryville, Emeryville, California
  - Satellite Dialysis Folsom, Folsom, California
  - Satellite Wellbound of Fremont, Fremont, California
  - Satellite Healthcare Gilroy, Gilroy, California
  - Satellite Healthcare Larkspur, Greenbrae, California
  - Satellite Healthcare Laguna Hills, Laguna Hills, California
  - Satellite Healthcare Merced, Merced, California
  - Satellite WellBound of Milpitas, Milpitas, California
  - Satellite WellBound of Modesto, Modesto, California
  - Satellite WellBound of North Modesto, Modesto, California
  - Satellite WellBound of Mountain View, Mountain View, California
  - Satellite Healthcare Orange, Orange, California
  - Satellite WellBound of Sacramento, Sacramento, California
  - Satellite WellBound of Sacramento University, Sacramento, California
  - Satellite Healthcare Sacramento, Sacramento, California
  - Satellite Healthcare San Carlos, San Carlos, California
  - Satellite WellBound of San Francisco, San Francisco, California
  - Satellite WellBound of San Jose, San Jose, California
  - Satellite WellBound of San Leandro, San Leandro, California
  - Satellite WellBound of San Mateo, San Mateo, California
  - Satellite WellBound of Santa Cruz, Santa Cruz, California
  - Satellite WellBound of Santa Rosa, Santa Rosa, California
  - Satellite Healthcare South Gate, South Gate, California
  - Satellite WellBound of Stockton, Stockton, California
  - Satellite Healthcare Tracy, Tracy, California
  - Satellite Healthcare Turlock West, Turlock, California
  - Satellite WellBound of Vallejo, Vallejo, California
  - Satellite Wellbound of Memphis, Memphis, Tennessee
  - Satellite WellBound of South Austin, Austin, Texas
  - Satellite WellBound of Austin, Austin, Texas
  - Satellite Healthcare Laredo South, Laredo, Texas

IPD SHARING:
Plan to Share IPD: Undecided
A de-identified data set of responses will be shared with the Kidney Research Institute at the University of Washington.